CLINICAL TRIAL: NCT01550523
Title: Phase 1 Study in Humans Evaluating the Safety of Rectus Sheath Implantation of Diffusion Chambers Encapsulating Autologous Malignant Glioma Cells Treated With Insulin-Like Growth Factor Receptor-1 Antisense Oligodeoxynucleotide in 12 Patients With Recurrent Malignant Glioma
Brief Title: Pilot Immunotherapy Trial for Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11G.532; JT 1587 (Other: JeffTrial Number)
Record Dates: First submitted 2012-02-14; First posted 2012-03-12 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Malignant Glioma of Brain
Keywords: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18-mer oligodeoxynucleotide (Experimental)
  Interventions: Drug: IGF-1R/AS ODN; Device: biodiffusion chamber

INTERVENTIONS:
Drug: IGF-1R/AS ODN — Patients will receive approximately 10 to 20 million IGF-1R/AS ODN treated tumor cells, encapsulated in diffusion chambers (maximum of 10), and re-implanted in the patient's abdomen within 24 hours after the surgery for a 24 hour period.
  Other Names: Nobel Sequence; Antisense; AS ODN
Device: biodiffusion chamber — The biodiffusion chamber is a simple construct comprised of two Lucite rings sealed on either side with a 0.1u mesh filter (Durapore, the Millipore Corporation). Autologous tumor cells pretreated with the IGF-1R AS ODN and resuspended with 2ug of exogenous IGF-1R AS ODN are added to the chamber. Implantation of the chambers (maximum 10 chambers) occurs 24 hours post surgery for 24 hours.

SUMMARY:
This human Phase I trial involves taking the patient's own tumor cells during surgical craniotomy, treating them with an investigational new drug (an antisense molecule) designed to shut down a targeted surface receptor protein, and re-implanting the cells, now encapsulated in small diffusion chambers the size of a dime in the patient's abdomen within 24 hours after the surgery. Loss of the surface receptor causes the tumor cells to die in a process called apoptosis. As the tumor cells die, they release small particles called exosomes, each full of tumor antigens. It is believed that these exosomes as well as the presence of the antisense molecule work together to activate the immune system against the tumor as they slowly diffuse out of the chamber. This combination product therefore serves as a slow-release antigen depot. Immune cells are immediately available for activation outside of the chamber because a wound was created to implant these tumor cells and a foreign body (the chamber) is present in the wound. The wound and the chamber fortify the initial immune response which eventually leads to the activation of immune system T cells that attack and eliminate the tumor. By training the immune system to recognize the tumor, the patient is also protected through immune surveillance from later tumor growth should the tumor recur. Compared to the other immunotherapy strategies, this treatment marshalls the native immune system (specifically the antigen presenting cells, or dendritic cells) rather than engineering the differentiation of these immune cells and re-injecting them. Compared to traditional treatment alternatives for tumor recurrence, including a boost of further radiation and more chemotherapy, this treatment represents potentially greater benefit with fewer risks.

This combination product serves as a therapeutic vaccine with an acceptable safety profile, which activates an anti-tumor adaptive immune response resulting in radiographic tumor regression.

DETAILED DESCRIPTION:
This trial will be an adaptation and continuation of a previously published trial, reproducing the original study size of 12 patients. Modifications from the previous trial include a modified oligodeoxynucleotide sequence and treatment at initial diagnosis, which would occur with concomitant standard therapy in an additional Phase 1 trial as a continuation if no rate-limiting toxicity is noted in the original Phase 1 arm. For practical purposes, a standard Phase 1 dose-escalation study is not possible with the current paradigm. Although we may have identified a distinct bioactive byproduct of IGF-1R/AS ODN-induced tumor cell apoptosis (exosomes), it is difficult to perform a dose escalation in a typical fashion. Also, antigen concentration can affect immune response in a biphasic manner: too little or too much can dampen an immune response, so even if the antigen or antigens were known, a typical pharmacologic dose escalation would not follow typical pharmacokinetics. For these reasons, we have designed a follow-on Phase 1 arm in which 32 patients will have therapy at initial surgery in 4 cohorts of 8 patients each. We will vary chamber number and implantation duration for each of the four cohorts in the additional Phase 1 arm. When we documented an increase in tumor infiltrating lymphocytes after treatment in our original trial, this observation provided preliminary supporting evidence that this therapeutic vaccine will elicit an adaptive immune response. We have designed the Phase 1 arm to further elucidate an immune response with a quantitative assessment of tumor specific T cells as well as circulating M2 macrophages before and after treatment. The design of the Phase 1 phase of the trial will allow a statistical analysis of both antigen dose (number of chambers) and time of exposure (chamber dwell time) as either variable may relate to any toxicity or treatment response.

A summary of the treatment paradigm includes: Pre-operative plasma leukopheresis, then surgery with tissue harvest and implantation of up to 10 chambers in the rectus sheath with IGF-1R/AS ODN as previously reported within 24 hours of craniotomy plus one chamber containing only phosphate buffered saline. Twelve patients treated for recurrent disease will be assessed for safety of the treatment. If the safety profile is acceptable, the trial will be followed by accrual of 32 patients in an additional Phase 1 trial as a continuation over approximately 3 years prospectively from Thomas Jefferson University Hospital and the Jefferson Hospital for Neuroscience. All patients who meet the eligibility criteria and agree to participate in this study will be potential candidates for therapy.

Pre-Operative Preparation - Patients will consent to a plasma leukopheresis at least 3 days prior to elective craniotomy. The PBMC will be stored for subsequent analysis of T cell responses, the presence of IL-10-producing M2 macrophages, and dendritic cell (DC) preparation. ELISPOT assays will be performed to measure T cell responses to autologous tumor cells and allogeneic tumor cells (U118 tumor lysate) utilizing cross-primed DC to assess both native anti-glioma immunity any acquired immunity after treatment. If U118 allogeneic glioma cells elicit a CTL response, this cell line may serve as an antigen source for future serial vaccination protocols.

A pre-operative PET scan as a baseline against which we can compare post-treatment PET scans as indicated.

Surgery and Tumor Cell Retrieval - Craniotomy and MRI-based image guided tumor resection will be performed on all study patients by an experienced neurosurgeon . All tested malignant gliomas obtained from craniotomies performed at Thomas Jefferson University have expressed the IGF-1R (M. Resnicoff, personal communication). During resection, viable tumor tissue will be confirmed by pathologic examination of frozen sections, and then sent to a BL-2 facility for disaggregation and plating in culture. Permanent section analysis will include an IGF-1R immunostain to determine the presence of IGF-1R. Once the cells are attached, cells will immediately be treated with IGF-1R/AS ODN. Tumor cells will be incubated with IGF-1R/AS ODN for a maximum of 6 hours and 106 cells will be then be loaded into each chamber and a target maximum of 10 chambers prepared. For all combination lot productions, two additional irradiated chambers and 300 ul of treated autologous tumor cells will be sent to microbiology for assessment of sterility according to FDA requirements. Greater than 5 and less than 10 chambers will be scored as a minor protocol violation. Recovery of no viable cells will be grounds for disenrollment from the protocol. Prior to implantation, the chambers will be irradiated with 5 Gy of X-irradiation as previously described. An additional tumor sample will be flash-frozen for exploratory research objectives. At the time of craniotomy the surgeon will create an abdominal acceptor site for subsequent diffusion chamber implantation in the rectus sheath. This implantation site was chosen for the following reasons: (1) it yielded objective favorable biological responses in the prior human Phase 1 trial; (2) this site will easily accommodate multiple chamber implantations; (3) this site should elicit a strong host response due to the extent of the wound, the introduction of a foreign body and its contents, the vasculature of the rectus sheath and muscle, and the favorable inguinal node lymphatic drainage from this site; and (4) exposure of the rectus sheath and muscle is familiar to neurosurgeons all of whom commonly perform ventricular-peritoneal shunts.

Biodiffusion Chamber Implantation/Explantation - Autologous tumor cell preparation, encapsulation in the biodiffusion chambers, irradiation, and chamber implantation/explantation are all procedures detailed in the Standard Operating Procedures Manual for IND #14379 (SOP 001). Briefly, at bedside in the intensive care unit the patient is sedated with intravenous Midazolam (Versed, 0.05 mg/kg repeated every 2 - 3 minutes to adequate sedation up to a maximum dose of 0.2mg/kg) and and Fentanyl (Sublimaze, 5mg which may be repeated every 5 minutes to a maximum dose of 20mg) and the wound infiltrated with up to 30 cc of 0.5% bupivicaine. With appropriate local anesthesia and sedation, the wound prepared at surgery is re-opened through the rectus sheath and up to 10 chambers are implanted between the rectus sheath and rectus muscle. The sheath is then re-approximated with 2-0 vicryl sutures and the skin re-approximated with 3-0 nylon sutures.The 24 hour period of implantation was chosen based on the favorable safety profile and promising biological responses noted in the previous human Phase 1 trial. Explantation involves the same process the following day with chamber explantation and a four layer wound closure.

Follow-up MRI imaging schedule The MRI studies at days 28 and 56 are acknowledged as not being done as standard of care because they would not reflect meaningful clinical data if patients received only standard of care treatment. The first surveillance MRIs are usually obtained around 3 months after surgery or other interventions such as radiation or chemotherapy. After this experimental treatment, however, we anticipate radiographic responses much earlier as documented in the prior human trial. In the prior trial, partial or complete radiographic responses were documented anywhere from 2 to 27 weeks after treatment. We interpret these early responses to be a reflection of an immune-mediated biological response.

Follow-up PET imaging schedule PET scans are scheduled at the discretion of the investigator to confirm disease progression.

Retreatment of Subjects will be considered for an anticipated subgroup of subjects initially participating in this protocol who have demonstrated immunocompetent responses associated with objective clinical and radiographic improvements after induction vaccination. Specifically, if serial assessments of T cell numbers and associated inflammatory cytokines, interferon, the INF-responsive cytokines CXCL9, CXCL10, and interleukin 6 are significantly elevated and associated with clinical and radiographic improvement.

Subjects entering the retreatment phase of the protocol will follow the same treatment plan with the exception of pre-operative plasma leukopheresis. Plasma leukopheresis previously collected will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Failure after previous standard of care initial treatment of glioblastoma multiforme.
* Documentation by MRI of an interval increase in nodular gadolinium enhancement consistent with recurrent malignant glioma suitable for therapeutic re-resection.
* Previous pathological diagnosis of WHO Grade IV glioma.
* All previous treatment interventions are acceptable.
* Patients must have an ECOG (Eastern Cooperative Oncology Group) performance status of 0, 1, or 2 or a KPS (Karnofsky Performance Score) of at least 60.
* Patients must be 18 years of age or older.
* Patients must sign an approved informed consent.
* Hemodynamically stable, consistent with Standard of Care values for patients undergoing elective tumor resection.

Exclusion Criteria:

* Females who are pregnant, nursing, or not inclined to use adequate contraceptive methods if necessary to prevent pregnancy during the study.
* An active second primary malignancy with the exception of basal cell or squamous cell skin carcinoma.
* Major concomitant medical illness inclusive of severe chronic obstructive pulmonary disease, symptomatic coronary artery disease, heart failure, recent major cerebrovascular accident, brittle diabetes, renal dialysis, end stage liver disease, or labile hypertension.
* Patients who have a history of heparin-induced thrombocytopenia or hypersensitivity to heparin, enoxaparin, or pork products.
* Patients with an abnormal INR (International Normalized Ratio of greater than 1.3), if repeatable and refractory to correction by routine methods.
* Patients who have documented deep venous thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02-09 (Actual); Primary Completion 2013-06-25 (Actual); Study Completion 2013-06-25 (Actual)

PRIMARY OUTCOMES:
To establish the safety profile of a combination product with an optimized Good Manufacturing Practices AS ODN in the treatment of patients with recurrent malignant glioma with concomitant assessment of any therapeutic impact. | Continuous throughout 24 month study participation.

SECONDARY OUTCOMES:
MRI based radiographic responses to treatment | <3 days prior to craniotomy, Day 28 post craniotomy, Day 56 post craniotomy, then every 3 months until 24 months (study completion at 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: David W Andrews, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital; Jefferson Hospital for Neurosciences, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Andrews DW, Resnicoff M, Flanders AE, Kenyon L, Curtis M, Merli G, Baserga R, Iliakis G, Aiken RD. Results of a pilot study involving the use of an antisense oligodeoxynucleotide directed against the insulin-like growth factor type I receptor in malignant astrocytomas. J Clin Oncol. 2001 Apr 15;19(8):2189-200. doi: 10.1200/JCO.2001.19.8.2189. PMID 11304771
- [Background] Agnelli G, Piovella F, Buoncristiani P, Severi P, Pini M, D'Angelo A, Beltrametti C, Damiani M, Andrioli GC, Pugliese R, Iorio A, Brambilla G. Enoxaparin plus compression stockings compared with compression stockings alone in the prevention of venous thromboembolism after elective neurosurgery. N Engl J Med. 1998 Jul 9;339(2):80-5. doi: 10.1056/NEJM199807093390204. PMID 9654538
- [Background] Agnelli G, Prandoni P, Santamaria MG, Bagatella P, Iorio A, Bazzan M, Moia M, Guazzaloca G, Bertoldi A, Tomasi C, Scannapieco G, Ageno W; Warfarin Optimal Duration Italian Trial Investigators. Three months versus one year of oral anticoagulant therapy for idiopathic deep venous thrombosis. Warfarin Optimal Duration Italian Trial Investigators. N Engl J Med. 2001 Jul 19;345(3):165-9. doi: 10.1056/NEJM200107193450302. PMID 11463010
- [Background] Baserga R. The insulin-like growth factor I receptor: a key to tumor growth? Cancer Res. 1995 Jan 15;55(2):249-52. PMID 7812953
- [Background] Brandes AA, Scelzi E, Salmistraro G, Ermani M, Carollo C, Berti F, Zampieri P, Baiocchi C, Fiorentino MV. Incidence of risk of thromboembolism during treatment high-grade gliomas: a prospective study. Eur J Cancer. 1997 Sep;33(10):1592-6. doi: 10.1016/s0959-8049(97)00167-6. PMID 9389920
- [Background] Cage TA, Lamborn KR, Ware ML, Frankfurt A, Chakalian L, Berger MS, McDermott MW. Adjuvant enoxaparin therapy may decrease the incidence of postoperative thrombotic events though does not increase the incidence of postoperative intracranial hemorrhage in patients with meningiomas. J Neurooncol. 2009 May;93(1):151-6. doi: 10.1007/s11060-009-9886-4. Epub 2009 May 9. PMID 19430892
- [Background] Carpentier A, Laigle-Donadey F, Zohar S, Capelle L, Behin A, Tibi A, Martin-Duverneuil N, Sanson M, Lacomblez L, Taillibert S, Puybasset L, Van Effenterre R, Delattre JY, Carpentier AF. Phase 1 trial of a CpG oligodeoxynucleotide for patients with recurrent glioblastoma. Neuro Oncol. 2006 Jan;8(1):60-6. doi: 10.1215/S1522851705000475. PMID 16443949
- [Background] Chaput N, Schartz NE, Andre F, Taieb J, Novault S, Bonnaventure P, Aubert N, Bernard J, Lemonnier F, Merad M, Adema G, Adams M, Ferrantini M, Carpentier AF, Escudier B, Tursz T, Angevin E, Zitvogel L. Exosomes as potent cell-free peptide-based vaccine. II. Exosomes in CpG adjuvants efficiently prime naive Tc1 lymphocytes leading to tumor rejection. J Immunol. 2004 Feb 15;172(4):2137-46. doi: 10.4049/jimmunol.172.4.2137. PMID 14764679
- [Background] Cosaceanu D, Carapancea M, Alexandru O, Budiu R, Martinsson HS, Starborg M, Vrabete M, Kanter L, Lewensohn R, Dricu A. Comparison of three approaches for inhibiting insulin-like growth factor I receptor and their effects on NSCLC cell lines in vitro. Growth Factors. 2007 Feb;25(1):1-8. doi: 10.1080/08977190600702865. PMID 17454144
- [Background] Cunningham CC, Holmlund JT, Schiller JH, Geary RS, Kwoh TJ, Dorr A, Nemunaitis J. A phase I trial of c-Raf kinase antisense oligonucleotide ISIS 5132 administered as a continuous intravenous infusion in patients with advanced cancer. Clin Cancer Res. 2000 May;6(5):1626-31. PMID 10815879
- [Background] Davidson A, Diamond B. Autoimmune diseases. N Engl J Med. 2001 Aug 2;345(5):340-50. doi: 10.1056/NEJM200108023450506. No abstract available. PMID 11484692
- [Background] Tang J, Flomenberg P, Harshyne L, Kenyon L, Andrews DW. Glioblastoma patients exhibit circulating tumor-specific CD8+ T cells. Clin Cancer Res. 2005 Jul 15;11(14):5292-9. doi: 10.1158/1078-0432.CCR-05-0545. PMID 16033848
- [Background] Tetri S, Hakala J, Juvela S, Saloheimo P, Pyhtinen J, Rusanen H, Savolainen ER, Hillbom M. Safety of low-dose subcutaneous enoxaparin for the prevention of venous thromboembolism after primary intracerebral haemorrhage. Thromb Res. 2008;123(2):206-12. doi: 10.1016/j.thromres.2008.01.018. Epub 2008 Apr 16. PMID 18420258
- [Background] Zimmerman RA. Imaging of adult central nervous system primary malignant gliomas. Staging and follow-up. Cancer. 1991 Feb 15;67(4 Suppl):1278-83. doi: 10.1002/1097-0142(19910215)67:4+3.0.co;2-u. PMID 1991289
- [Background] Dorn A, Kippenberger S. Clinical application of CpG-, non-CpG-, and antisense oligodeoxynucleotides as immunomodulators. Curr Opin Mol Ther. 2008 Feb;10(1):10-20. PMID 18228177